CLINICAL TRIAL: NCT02223533
Title: Multimodal Analgesia With Interfascial Continuous Wound Infiltration of a Local Anaesthetic vs Intravenous Opioids After Laparoscopic Colon Surgery: A Randomized Clinical Trial.
Brief Title: Multimodal Analgesia With Interfascial Continuous Wound Infiltration: A Randomized Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Galdakao-Usansolo (Other Government)
Responsible Party: Principal Investigator, Sorkunde Telletxea, MD, PhD, MD, PhD, Hospital Galdakao-Usansolo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sork-2011111058
Record Dates: First submitted 2014-08-18; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Pain
Keywords: analgesia; post-operative; wound catheter infusion; laparoscopic colon surgery
MeSH Terms: conditions — Pain; Agnosia | interventions — Morphine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wound catheter (Experimental): analgesia with wound catheter after colon surgery
  Interventions: Device: 19Gx500-mm Pajunk InfiltraLong® catheter
- morphine (Active Comparator): analgesia with morphine after colon surgery
  Interventions: Drug: morphine

INTERVENTIONS:
Device: 19Gx500-mm Pajunk InfiltraLong® catheter — Before completing the surgery, the surgical team inserted a 19Gx500-mm Pajunk InfiltraLong® catheter with multiple perforations in the last few centimeters before the tip to allow for local anesthetic administration.
  Arms: Wound catheter
Drug: morphine — After the intervention patients had access to intravenous morphine via a patient-controlled analgesia
  Arms: morphine

SUMMARY:
Objectives: For major laparoscopic surgery, as with open surgery a multimodal analgesia plan can help control postoperative pain. Placing a wound catheter intraoperatively following colon surgery could optimize the control of acute pain with less consumption of opioids and few adverse effects.

Methods: We conducted a prospective, randomized, study of 103 patients scheduled to undergo laparoscopic colon surgery for cancer in Galdakao-Usansolo Hospital.

Patients were recruited and randomly allocated to wound catheter placement plus standard postoperative analgesia or standard postoperative analgesia alone. A physician from the acute pain management unit monitored all patients for at multiple points over the first 48 hours after surgery. The primary outcome variables were verbal numeric pain scale (NRS) scores and amount of intravenous morphine used via patient controlled infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for the study if they were aged 18 years or older, with an American Society of Anesthesiologists (ASA) 14 grade of I to IV (anaesthetic risk), were scheduled to undergo laparoscopic colon surgery, and voluntarily agreed to participate by signing an informed consent form.

Exclusion Criteria:

* Patients were excluded if they were allergic to amides or pyrazolones, were likely to require conversion to open surgery with laparotomy, were long-term users of opioids, required emergency surgery, were unable to participate due to cognitive deterioration, or declined to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Numerical Rating Pain Scale (NRS) after laparoscopic colon surgery using interfascial continuous wound infiltration | Over the 48 hours after laparoscopic colon surgery
  Numerical Rating Pain Scale was used to measure the after-intervention Pain. This scale is widely used and shows good correlation with the Visual Analogue scale, specifically in the case of elderly individuals. Compared to other scales, it has low error rates and high validity. This score was assessed in all the participants.
Assessment of intravenous morphine consumption after laparoscopic colon surgery | Over the 48 hours after laparoscopic colon surgery
  Intravenous morphine consumption was administrated via patient-controlled analgesia device. The consumption was evaluated in all participants in the study at the following measurement points: at 30 min, 2h, 8h, 24h, and 48h after the intervention.

SECONDARY OUTCOMES:
Complications related to intravenous morphine consumption | Over the 48 hours after laparoscopic colon surgery
  Complications related to intravenous morphine consumption were measured: nausea, vomiting and pruritus throughout the treatment period. Paralytic ileus awas measured 24h after surgery. This was assessed for all patients. Moreover, especially for patients belonging to the experimental group, potential adverse effects from placement of the wound catheter such as infection or haematoma at the surgical site or potential toxicity of local anesthetic (e.g., tinnitus, obnubilation) were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sorkunde Telletxea, MD, PhD, Principal Investigator — Hospital Galdakao-Usansolo
Locations (1):
- Hospital de GAldakao-Usansolo, Usansolo, Biscay, Spain